CLINICAL TRIAL: NCT03763773
Title: Prediction of Outcomes With a Miniaturized Transesophageal Echocardiography Probe in Patients With Acute Respiratory Distress Syndrome
Acronym: PreMiTE-ARDS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_30; 2018-A01463-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: respiratory variations,; superior vena cava; prognosis.
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Superior Vena cava Respiratory Collapse Index (cVCS) is a haemodynamic parameter measured exclusively by transoesophageal ultrasound (TEE), which is used to assess cardiac precharge-dependence status. This may be an important prognostic factor in ARDS because it is a sign of hypervolemia and right heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in Resuscitation, Emergency or Intensive Care Units at the Roger Salengro Hospital at Lille University Hospital.
* With acute respiratory distress syndrome of intermediate or severe severity (1) for less than 24 hours.
* Mechanical ventilation with tracheal intubation or tracheostomy, in controlled assisted ventilation (VAC) mode.
* Patient adapted to mechanical ventilation (no triggering of spontaneous ventilation cycle in VAC mode verified by the equality between the respiratory rate prescribed on the ventilator and the actual respiratory rate of the patient).

Exclusion Criteria:

* Patient under extracorporeal respiratory assistance at the time of inclusion.
* Anomalies or pathologies that make it dangerous or impossible to introduce an ETO probe:

  * Fistula, perforation, stenosis, varicose vein or diverticulum of the esophagus and / or stomach
  * History of esophageal and / or gastric surgery
  * Caustic lesions of the esophagus and / stomach
  * Tumor or history of oropharyngeal surgery
  * Unstable lesions of the cervical spine
  * Coagulopathy (thrombocytopenia <50 109 / L and / or TP <50%).
* Impossibility of measuring the diameter of the superior vena cava and cVCS in ETO due to poor echogenicity.
* Pregnant woman.
* Therapeutic limitation measures limiting the treatment of organ failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with mechanical ventilation hospitalized in intensive care, emergency or intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Number of days lived without mechanical ventilation | at 28 days
  This variable will be defined as follows:duration = 28 -x -y. where x is the number of days living under mechanical ventilation during the first 28 days and the number of days in the first 28 days.

SECONDARY OUTCOMES:
number of patient of death | At 28 days, at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Preau, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

REFERENCES:
- [Derived] Preau S, Pouly O, Ederkaoui M, Durand A, Bourel C, Onimus T, Cadart L, Labreuche J, Howsam M, Favory R, Pierre A. Lack of preload responsiveness may determine poor clinical outcomes in mechanically ventilated patients with ARDS. Crit Care. 2025 May 1;29(1):172. doi: 10.1186/s13054-025-05409-4. PMID 40312326